CLINICAL TRIAL: NCT06894589
Title: Assessment of the Perceptions and Opinions of Staff Working in Prisons and Detention Centers on the Use of Psychoactive Substances in Prisons and Harm Reduction
Brief Title: Assessment of the Perceptions and Opinions of Staff Working of Prisons and Detention Centers on the Use of Psychoactive Substances in Prisons and Harm Reduction (PERRCEP)
Acronym: PERRCEP
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0333 - PERRCEP
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-01

CONDITIONS: Harm Reduction; Prisoners
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation, through an anonymous questionnaire, of the perceptions and opinions of staff working in prisons and detention centers in Brittany regarding the consumption of illicit substances and harm reduction measures in prison environment. The secondary objective of the study will be to assess training needs and explore factors associated with better adherence to the implementation of harm reduction measures.

DETAILED DESCRIPTION:
A first contact will be made by email with the heads of institutions, directors of Penitentiary Rentegration Services), and coordinating doctors of healthcare units to inform them about the study's objectives and procedures, and to request their institution's and service's participation.

If they agree to participate, volunteer key contacts will be identified in each institution to relay the information to the staff working in the institution and ensure the distribution of the questionnaire.

The study's responsible doctor will meet with one of the resident investigators for a preliminary informational meeting with the institution's director, the SPIP director, and the identified key staff members. The questionnaires will be handed to the key contacts at that time.

A "non-opposition" letter will be individually distributed with each anonymous questionnaire to provide further details about the study for which their participation is requested.

After answering, participants will be able to place the questionnaire in the provided envelope, and then into a sealed ballot box.

After the answering period, the investigator will go back to prisons and detention centers to collect the ballot boxes.

The data from each paper questionnaire will be transcribed by the residents onto an online platform using the Lime Survey® software.

The statistician of UBO (university of Brest) will have access to the data on Lime Survey® in order to perform the statistical analyses as described below.

The statistician will make a descriptive analysis of the results and the an analytical study will research factors associated with improved adherence to harm reduction mesures : profession exercised; seniority; harm reduction training; age

ELIGIBILITY:
Inclusion Criteria:

* working person of remand center of Brest, Vannes, Rennes, Saint-Malo, Lorient and Saint-Brieuc, who has answered the questionnaire
* working person of detention center of Lorient and Rennes, who answered the questionnaire

Exclusion Criteria:

* person opposing participation in the study
* person under legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Working person of remand center of Brest, Vannes, Rennes, Saint-Malo, Lorient and Saint-Brieuc, and detention center of Lorient and Rennes :
  * healthcare staff, divided into 5 sectors : somatic, psychiatric, odontology, addictology, pharmacy)
  * prison warders
  * Reintegration support service (in french : Service pénitentiaire d'insertion et de probation)
  * other prison staff
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
perceptions and opinions of staff working in prisons and detention centers in Brittany regarding the consumption of illicit substances and harm reduction measures. | from january 2025 to may 2025
  descriptive analysis of the results

SECONDARY OUTCOMES:
Assess training needs and research factors associated with improved adherence to harm reduction mesures | from january 2025 to may 2025
  An analytical study will research factors associated with improved adherence to harm reduction mesures : profession exercised; seniority; harm reduction training; age.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement